CLINICAL TRIAL: NCT03846986
Title: Effect of Added Fruit Pomace Fiber and Whole Fruit on Postprandial Glycemia in Apple
Brief Title: Postprandial Glycemia in Apple Products
Acronym: PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2018-115
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Apple pomace fiber; Glycemic response; Apple

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apple Juice1 (Active Comparator): 100% Apple Juice
  Interventions: Dietary Supplement: Apple Juice1
- Apple Juice2 (Experimental): 100% Apple Juice with enzyme-treated apple pomace fiber
  Interventions: Dietary Supplement: Apple Juice2
- Raw Apple (Placebo Comparator): Raw Apple
  Interventions: Dietary Supplement: Raw Apple

INTERVENTIONS:
Dietary Supplement: Apple Juice1 — Apple Juice1
  Other Names: Apple Juice
  Arms: Apple Juice1
Dietary Supplement: Apple Juice2 — 100% Apple Juice with enzyme-treated apple pomace fiber
  Other Names: Apple Juice with Pomace Fiber
  Arms: Apple Juice2
Dietary Supplement: Raw Apple — Raw Apple
  Arms: Raw Apple

SUMMARY:
The primary objective of the study is to compare the effects of a whole apple, apple juice alone, and apple juice with pomace on 2 hr glycemic response as measured by maximal glucose concentration

DETAILED DESCRIPTION:
This study is a randomized, 3-arm, within subject cross-over trial allowing for three acute evaluations of 100% Apple Juice (235 g), 100% Apple Juice with enzyme-treated apple pomace fiber (129 g apple juice with 106 g apple pomace), and raw apple (230 g with skin edible portion - not including core or stem) on glucose and insulin responses in fifty-two healthy men and women aged 20-45 years.

A planned sample size of 70 will be enrolled into the study. This study will require one initial screening visit and 3 study visits. This study will take approximately 3-4 weeks per subject to complete.

The initial screening visit will take ~2 hours and provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, body composition measurement, vital signs, fasting blood glucose test (finger prick), a vein access scale evaluation, online 24-hr diet recall, and completion of a survey relate to general eating, health, and exercise habits. For women, a pregnancy test will be conducted.

If willing and eligible to participate, subjects will be invited to participate in the study for 3 study day visits. Eligible subjects will be instructed to follow a relatively low polyphenolic diet for at least 1-week prior the beginning of the study and continue for the duration of the study.

Each Study Day visit will last about ~3 hours. The day before each of the 3 Study Day visits, subjects will be asked to consume the same dinner meal and record on a food record. At each Study Day visit, subjects will arrive at the clinic after fasting for 10 to 12 hours and in a well-hydrated and well-rested state.

Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a Licensed Health Care Professional will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. Subjects will be randomized to receive one of study products based on randomized treatment sequences for 3 study visits immediately after fasting blood draw.

Participants will come to the research site on 3 separate occasions separated by a washout period. On each occasion 2 fasting blood samples will be obtained at 5 min intervals (-5, 0 minute (min)). Subjects will then consume one of the 3 treatments. Further blood samples will be taken at 15, 25, 30, 35, 40, 45, 60, 75, 90, 105 and 120 min. Self-reported visual analog scales (VAS) will be used to measure subject hunger, fullness, desire to eat, and prospective food intake at 0, 15, 30, 60, 90, and 120 min. After completion of all study procedures and data/sample collection for the day, the catheter will be removed and subjects will be evaluated for safety and/or discomfort/symptoms before leaving the study site. They will be given a take-home snack and given written instructions in preparation for the next visit. Study day visits will be scheduled at least 3 days apart but no more than 7 days.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is a male or female, 20-45 years of age, inclusive.

  * Subject has a BMI of 20.0-24.9 kg/m2, inclusive and weight ≥ 110 lb at screening visit.
  * Subject is willing to maintain his/her usual physical activity pattern throughout the study period.
  * Subject is willing to follow study instructions including compliance with dietary restrictions, consumption of study beverage, and study visit schedule.
  * Subject is judged to be in good health on the basis of the medical history.
  * Subject is willing to abstain from alcohol consumption for 24 hours prior to study visit.
  * Exercise to be maintained throughout study duration, including 3 days before study visit
  * Subject is willing to maintain stable dose of current vitamins, minerals, supplements and medications not interfering with study outcomes, including birth control, throughout study duration.
  * Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator/s and is willing to complete study procedures

Exclusion Criteria:

* •Subject has fasting finger prick glucose >100 mg/dL.

  * Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at the screening visit.
  * Subject has had major trauma or a surgical event within 2 months of study visit 1.
  * Subject has had a weight change ≥4.5 kg within 2 months of visit, taking weight loss drugs, or has had bariatric surgery or other weight reduction surgery (ie. liposuction, laser fat removal, etc)
  * Subject has a history or presence of clinically important endocrine, cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary, or gastrointestinal disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
  * Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
  * Subject has a history of extreme dietary habits, as judged by the Investigator (e.g., Atkins diet, etc.).
  * Subject has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
  * Subject has a known intolerance or sensitivity to any ingredients in the study products.
  * Subject has used medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, hypoglycemic medications, and systemic corticosteroids 2 weeks prior to visit 1 and throughout the study.
  * Subject taking systemic steroids, extreme alcohol use, or drug user.
  * Subject has vein access score less than 7
  * Subject is a female, who is pregnant, planning to be pregnant during the study period or lactating.
  * Subject is a current smoker. Past smoker abstinence for less than 2 years.
  * Subject has participated in any clinical trial within 30d prior to enrollment.
  * No participation in another Sponsored protocol within 6 months prior to enrollment

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose maximal concentration (Cmax) over 2 hours | Postprandial 2 hours
  Plasma Glucose maximal concentration (Cmax) over 2 hours

SECONDARY OUTCOMES:
Changes in Plasma Glucose concentration as measured by incremental area under the curve (iAUC) over 2 hours | Postprandial 2 hours
  Changes in plasma glucose concentration as measured by iAUC over a 2-hour Postprandial Test day after administration of active treatment compared to control treatment

OTHER OUTCOMES:
Time to plasma glucose maximal concentration (Tmax) over 2 hours | Postprandial 2 hours
  Time to plasma glucose maximal concentration (Tmax) over 2 hours
Plasma Insulin Cmax over 2 hours | Postprandial 2 hours
  Plasma Insulin Cmax over 2 hours
Changes in plasma insulin concentration as measured by iAUC over a 2-hour period Postprandial Test day after administration of active treatment compared to control treatment | Postprandial 2 hours
  Plasma Insulin iAUC over 2 hours
Time to Plasma Insulin Maximal concentration (Tmax) over 2 hour2 | Postprandial 2 hours
  Time to Plasma Insulin Maximal concentration (Tmax) over 2 hours
Changes in postprandial subjective satiety responses using visual analog scales (VAS) of Hunger over 2 hours | Postprandial 2 hours
  Self-reported Subjective VAS of Hunger by placing a marker (ranged in 0 to 100 mm) on the line scale anchored by opposing terms(eg. From Extremely to Not at all) at designated timepoints
Changes in postprandial subjective satiety responses using visual analog scales (VAS) of Fullness over 2 hours | Postprandial 2 hours
  Self-reported Subjective VAS of Fullness by placing a marker (ranged in 0 to 100 mm) on the line scale anchored by opposing terms (eg. From Extremely to Not at all) at designated timepoints
Changes in postprandial subjective satiety responses using visual analog scales (VAS) of desire to eat over 2 hours | Postprandial 2 hours
  Self-reported Subjective VAS of Desire to eat by placing a marker (ranged in 0 to 100 mm) on the line scale anchored by opposing terms (eg. From Extremely to Not at all) at designated timepoints
Changes in postprandial subjective satiety responses using visual analog scales (VAS) of Prospective food intake over 2 hours | Postprandial 2 hours
  Self-reported Subjective VAS of Prospective food intake by placing a marker (ranged in 0 to 100 mm) on the line scale anchored by opposing terms (eg. From Extremely to Not at all) at designated timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Study Chair — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No